CLINICAL TRIAL: NCT01514864
Title: Phase II Trial of Dasatinib in Subjects With Advanced Cancers Harboring DDR2 Mutation or Inactivating B-RAF Mutation
Brief Title: Trial of Dasatinib in Patients With Advanced Cancers Harboring DDR2 Mutation or Inactivating B-RAF Mutation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy and slow accrual
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-385; 2011-003128-11 (EudraCT Number)
Record Dates: First submitted 2012-01-18; First posted 2012-01-23 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Non-small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) (Experimental): Participants with nonsmall-cell lung cancer (NSCLC) and an inactivating B-RAF mutation received dasatinib, 140 mg, once daily as a tablet until unacceptable toxicity or disease progression occurred
  Interventions: Drug: Dasatinib
- Dasatinib, 140 mg (NSCLC With DDR2 Mutation) (Experimental): Participants with NSCLC and a discoidin domain receptor 2 (DDR2) mutation received dasatinib, 140 mg, once daily as a tablet until unacceptable toxicity or disease progression occurred
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablet, oral, 140 mg, once daily until unacceptable toxicity or disease progression

SUMMARY:
The purpose of this study is to establish whether patients with malignancy harboring a discoidin domain receptor 2 mutation or an inactivating B-RAF mutation will respond to dasatinib.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria

* Diagnosis of advanced malignancy, nonsmall-cell lung cancer (NSCLC) only during stage 1 of accrual.
* Nonsynonymous mutation of B-RAF or DDR2, defined as follows:.

  i) NSCLC with inactivating B-RAF mutation.

ii) NSCLC with discoidin domain receptor 2 (DDR2) mutation.

iii) Malignancy of other histology with DDR2 mutation or inactivating B-RAF mutation, or NSCLC having a B-RAF mutation that is not functionally characterized.

* At least 1 target lesion per Response Evaluation Criteria in Solid Tumors, vol 1.1, on baseline staging evaluation.
* Disease progression after ≥ 1 prior treatment regimen.

Exclusion Criteria

* Pleural or pericardial effusion, Grade >1.
* QTcF >470 msec (Grade ≥2) or diagnosed congenital long QT syndrome.
* Absolute granulocyte count <1500/mm^3.
* Hemoglobin level <10 g/dL.
* Platelet count < 75,000/mm^3.
* Serum calcium level <institutional lower limit of normal.
* Hypokalemia, hypophosphatemia, or hypomagnesemia, Grade >1, despite supplementation.
* Creatinine >3*institutional upper limit of normal (ULN).
* Total bilirubin level >1.5*ULN.
* Alanine transaminase level >3*ULN.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2014-07-23 (Actual); Study Completion 2014-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (3):
  - H. Lee Moffitt Cancer & Research Institute, Tampa, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, New York, New York
- Brazil (3):
  - Local Institution, Barretos, São Paulo
  - Local Institution, S?o Paulo, São Paulo
  - Local Institution, São Paulo
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada
- Germany (3):
  - Local Institution, Cologne
  - Local Institution, Frankfurt
  - Local Institution, Heidelberg
- Poland (3):
  - Local Institution, Gdansk
  - Local Institution, Lodz
  - Local Institution, Warsaw
- Local Institution, Taipei, Taiwan
- United Kingdom (7):
  - Local Institution, Cambridge, Cambridgeshire
  - Local Institution, London, Greater London
  - Local Institution, Manchester, Greater Manchester
  - Local Institution, Gwent, Gwent
  - Local Institution, Edinburgh, Midlothian
  - Local Institution, Sutton, Surrey
  - Local Institution, Cambridge

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 19 patients were enrolled, and 14 received treatment in 2 cohorts: 9 with nonsmall-cell lung cancer (NSCLC) and an inactivating B-RAF mutation and 5 with NSCLC and a discoidin domain receptor 2 (DDR2) mutation.
Period: Overall Study
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation)
Started | 9 | 5
Completed | 0 (Study was terminated; no patients completed study treatment) | 0
Not Completed | 9 | 5
Not completed — Disease progression | 7 | 5
Not completed — Study drug toxicity | 2 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation) | Total
Number analyzed (Participants) | 9 | 5 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 6 | 2 | 8
Age, Continuous [Median (Full Range); unit: Years] | 67.0 [51.0 to 75.0] | 63.0 [50.0 to 73.0] | 66.5 [50.0 to 75.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic/Latino | 1 | 0 | 1
  Not Hispanic/Latino | 5 | 5 | 10
  Not reported | 3 | 0 | 3
Time from cancer diagnosis to start of study therapy [Median (Full Range); unit: Months] | 14.4 [6.2 to 21.7] | 8.5 [1.5 to 51.6] | 12.1 [1.5 to 51.6]
Tumor Type [Number; unit: Participants]
  Nonsmall-cell lung carcinoma | 9 | 5 | 14
  Other | 0 | 0 | 0
Nonsmall-cell lung carcinoma histology [Number; unit: Participants]
  Adenocarcinoma | 7 | 1 | 8
  Bronco-alveolar carcinoma | 1 | 0 | 1
  Large cell carcinoma | 1 | 0 | 1
  Squamous cell carcinoma | 0 | 4 | 4
Histopathologic Grade [Number; unit: Participants]
  G2-moderately differentiated | 2 | 2 | 4
  G3-poorly differentiated | 2 | 0 | 2
  GX-grade cannot be assessed | 5 | 3 | 8
Baseline Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — ECOG is a 6-item scale used to assess disease progression, daily functioning, and appropriate treatment and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all predisease performance without restriction and (worst score) 5=death.
  Participants
    ECOG score 0 | 1 | 1 | 2
    ECOG score 1 | 6 | 3 | 9
    ECOG score 2 | 2 | 1 | 3
Number of Index Lesions [Number; unit: Participants]
  1 | 2 | 1 | 3
  2 | 0 | 2 | 2
  3 | 4 | 1 | 5
  4 | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of patients with best tumor response of either Partial Response (a 30% or greater decrease in the sum of the longest diameter [LD] of all lesions in reference to the baseline sum LD) or Complete Response (disappearance of clinical and radiologic evidence of target lesions), according to Response Evaluation Criteria in Solid Tumors.
Time Frame: From enrollment of last patient to 24 months or until all patients have died, whichever occurs first
Population: All participants who received at least 1 dose of study drug. Because no patients had a response of CR or PR, ORR could not be calculated.
Groups:
- Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation): Participants with nonsmall-cell lung cancer (NSCLC) with inactivating B-RAF mutation received dasatinib, 140 mg, once daily as a tablet until unacceptable toxicity or disease progression occurred
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first assessment documentation of partial response (PR) or complete response (CR) until the first assessment documentation of disease progression.
Time Frame: From enrollment of last patient to 24 months or until all patients have died, whichever occurs first
Population: All participants who received at least 1 dose of study drug. Because no patients had a response of CR or PR, DOR could not be calculated.
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment start date to the date of death. If a patient does not die, survival will be censored on the last date the patient was known to be alive.
Time Frame: From enrollment of last patient to 24 months or until all patients have died, whichever occurs first
Population: All participants who received treatment
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation)
Number analyzed (Participants) | 9 | 5
Months | 3.06 [0.76 to 6.47] | 4.21 [0.82 to NA] — The upper limit Confidence Interval cannot be estimated

4. Secondary Outcome: Progression-free Survival (PFS) Distribution
Description: PFS distribution is defined as the percentage of patients with no documentation of disease progression at a specified time point. Confidence interval computed using the Brookmeyer and Crowley method
Time Frame: From Day 1 of study treatment to Week 12
Population: All participants who received at least 1 dose of study drug
Measure: Median (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation)
Number analyzed (Participants) | 9 | 5
Percentage of participants | 1.41 [0.72 to 1.87] | 1.38 [0.59 to 2.96]

5. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from treatment start date to the earliest evidence of disease progression or death. Patients who die or whose disease does not progress will be censored on the date of their last tumor assessment.
Time Frame: From Day 1 of study treatment to Week 12
Population: All participants who received at least 1 dose of study drug
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation)
Number analyzed (Participants) | 9 | 5
Months | 1.41 [0.72 to 1.87] | 1.38 [0.59 to 2.96]

6. Secondary Outcome: Number of Patients With Death as Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, Adverse Events (AEs) Leading to Discontinuation, and Drug-related AEs Leading to Discontinuation
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=having certain, probable, possible, or unknown relationship to study drug.
Time Frame: From enrollment of last patient to 24 months or until all patients have died, whichever occurs first
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Dasatinib, 140 mg (NSCLC With Inactivating B-RAF Mutation) | Dasatinib, 140 mg (NSCLC With DDR2 Mutation)
Number analyzed (Participants) | 9 | 5
Participants
  Death | 8 | 4
  Death within 30 days of last treatment | 3 | 1
  SAEs | 7 | 4
  Drug-related SAEs | 0 | 1
  AEs leading to discontinuation | 7 | 2
  Drug-related AEs leading to discontinuation | 2 | 0
  Drug-related AEs | 6 | 3

7. Secondary Outcome: Number of Participants With Laboratory Testing Results That Meet the Criteria for Grade 3 or 4 Abnormality
Description: Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living. Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living. Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to adverse event. Laboratory values graded by Common Terminology Criteria for Adverse Events, volume 3. Hemoglobin, Grade 3: <8.0 - 6.5 g/dL, <4.9-4.0 mmol/L, <80-65 g/L. Alkaline phosphatase, Grade 3: >5.0-20.0*upper limit of normal (ULN). Total bilirubin, Grade 3: >3.0-10.0*ULN. Calcium, low, Grade 3: <7.0-6.0 mg/dL, <1.75-1.5 mmol/L.
Time Frame: From enrollment of last patient to 24 months or until all patients have died, whichever occurs first
Population: All participants who received study drug.
Measure: Number; unit: Participants
Groups:
- Dasatinib, 140 mg: Participants with nonsmall-cell lung cancer (NSCLC) received dasatinib, 140 mg, once daily as a tablet until unacceptable toxicity or disease progression occurred. Data from both arms were combined for safety reporting, because the safety profile of dasatinib should not have be affected by the type of mutation in the tumor. In addition, pooling the data from both arms increased the robustness of the data set.
Arm/Group | Dasatinib, 140 mg
Number analyzed (Participants) | 14
Participants
  Hemoglobin, Grade 3 | 2
  Alkaline phosphatase, Grade 3 | 1
  Total bilirubin, Grade 3 | 1
  Calcium, low, Grade 3 | 1

ADVERSE EVENTS:
Groups:
- Dasatinib, 140 mg: Participants with nonsmall-cell lung cancer received dasatinib, 140 mg, once daily as a tablet until unacceptable toxicity or disease progression occurred. Data from both arms were combined for safety reporting, because the safety profile of dasatinib should not have be affected by the type of mutation in the tumor. In addition, pooling the data from both arms increased the robustness of the data set.
Arm/Group | Dasatinib, 140 mg
Serious Adverse Events (participants affected / at risk) | 11/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 140 mg (N=14)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
General physical health deterioration (General disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Angina unstable (Cardiac disorders) | 1
Haemoglobin decreased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Lipase increased (Investigations) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain (General disorders) | 1
Panic reaction (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib, 140 mg (N=14)
Blood alkaline phosphatase increased (Investigations) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Hepatic pain (Hepatobiliary disorders) | 1
Pyrexia (General disorders) | 2
Sedation (Nervous system disorders) | 1
Uveitis (Eye disorders) | 1
Calcium ionised increased (Investigations) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Eyelid oedema (Eye disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Vision blurred (Eye disorders) | 1
Blood alkaline phosphatase (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Deep vein thrombosis (Vascular disorders) | 1
Fatigue (General disorders) | 7
Headache (Nervous system disorders) | 3
Lower respiratory tract infection (Infections and infestations) | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Anxiety (Psychiatric disorders) | 2
Asthenia (General disorders) | 1
Blood glucose increased (Investigations) | 1
Confusional state (Psychiatric disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Oedema peripheral (General disorders) | 3
Parosmia (Nervous system disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Vasculitis (Vascular disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Blood albumin decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Oedema (General disorders) | 2
Pneumonia (Infections and infestations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Viral infection (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Extravasation (General disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Lipase increased (Investigations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain (General disorders) | 2
Electrocardiogram ST segment elevation (Investigations) | 1
Eye disorder (Eye disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Pain (General disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Urinary straining (Renal and urinary disorders) | 1
Chills (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Insomnia (Psychiatric disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Weight decreased (Investigations) | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of efficacy and slow enrollment of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.